CLINICAL TRIAL: NCT07300865
Title: Does the Thickness of the Gastrostomy Affect the Incidence of Complications? A Prospective Randomized Single-Center Study in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Therese Hössjer (Other)
Collaborators: Uppsala University (Other); Uppsala University Hospital (Other)
Responsible Party: Sponsor-Investigator, Therese Hössjer, Pediatric Surgeon, PhD-student, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-03305-01
Record Dates: First submitted 2025-12-20; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Gastrostomy Complications; Gastrostomy Size; Food Intolerance; Granuloma
Keywords: laparoscopic gastrostomy; complications; pediatric surgery; children; granuloma
MeSH Terms: conditions — Food Intolerance; Granuloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Children recieving 12 Fr gastrostomy tube (Other)
  Interventions: Device: 12 Fr gastrostomy tube/button
- Children recieving 14 Fr gastrostomy tube (Other)
  Interventions: Device: 14 Fr gastrostomy tube/button

INTERVENTIONS:
Device: 12 Fr gastrostomy tube/button — Patients in this arm will recieve 12 Fr size gastrostomy tube/ button
  Other Names: 12 Fr
  Arms: Children recieving 12 Fr gastrostomy tube
Device: 14 Fr gastrostomy tube/button — Patients in this arm will recieve 14 Fr size gastrostomy tube/ button
  Other Names: 14 Fr
  Arms: Children recieving 14 Fr gastrostomy tube

SUMMARY:
The goal of this interventional study is to compare two different sizes of a gastrostomy tube in children and the incidence of complications three months postoperatively. The study is questionnare-based and both the family and health care personel will fill in the formula about complications at the re-visit when the tube is changed the first time at three months postoperatively. Complications requested are: granuloma, infection, pain, dislocation and leakage.

DETAILED DESCRIPTION:
Project plan Does gastrostomy tube thickness affect incidence of complications?

Hypothesis A 12 Fr gastrostomy tube is associated with fewer complications than a 14 Fr tube.

Aim To investigate if the rate of postoperative complications is reduced when a 12 Fr gastrostomy is used instead of a 14 Fr.

Overview Placement of a gastrostomy is indicated in children with long term need of enteral nutrition where oral intake is inadequate and there is at least a partially functioning digestive tract [1]. The operative procedure includes creation of a channel through the stomach- and abdominal wall with placement of a tube. The tube keeps the channel open and enables feeding of and medication to the patient. There are different ways of establishing a gastrostomy: laparoscopic, percutaneous, radiologically assisted and open techniques. Some researchers consider the laparoscopic approach to be the most preferable and safe option while others prefer the percutaneous or open technique [2,3,4,5].

In Sweden approximately 300-400 children (0-18 years) receive a gastrostomy yearly, and it is one of the most common inpatient care interventions in children. The majority of patients have an underlying neurological disease with multiple somatic and/or cognitive impairments. Other indications include failure to thrive, nausea during cancer treatment, metabolic disorders, and gastrointestinal failure [6].

For most of the children and families the gastrostomy facilitates their everyday life and improve their well-being. Unfortunately, gastrostomies are associated with several minor complications which cause repeated contacts with healthcare providers in this already vulnerable patient group. Common complications are granuloma, infection, leakage, pain and dislocation, where granulomas are as common as 42-60% [3,4,7]. A granuloma, or granulation tissue, is formed in response to inflammation or a wound. It is a type of vascular connective tissue consisting of lymphoid cells, macrophages and plasma cells, which bleeds easily and produces exudate [8].

Today there is a lack of evidence on what size of gastrostomies should be used. Most commonly used thicknesses are 12 Fr and 14 Fr. One retrospective study showed that a 12 Fr gastrostomy tube were four times as likely to dislocate, than a 14 Fr gastrostomy [9]. In a previously published observational study we could not see that relation [10]. Instead, we found that a 12 Fr tube seems to be associated with fewer complications than other thicknesses. Since data seems to disperse, we aim to conduct this prospective randomised single-centre study to find out whether a 12 Fr tube thickness can reduce post-operative complications after gastrostomy compared to a 14 Fr.

Method

All children 0-15 years planned for a gastrostomy at Dep Pediatric Surgery in Uppsala will be invited to the study. After oral and written information, patient or caregivers will be asked to sign the form of consent. On the day of operation, the patient will be randomized to either 12 Fr or 14 Fr tube size of the gastrostomy. The surgeon will fill in the tube size in a questionary presented in appendix 2.1.

After three months the gastrostomy button should be changed to a new one, according to National guidelines for gastrostomies, which is done as an out patient visit at a nurse. Questionaries, including information about complications, will be filled out both by the nurse and the patient or caregivers.

The information from the three questionaries will be stored by the principal researcher at each clinic, and deidentified data will be filled out in an excel-file. The main researcher and doctoral student will then compile the data and perform statistical analyses. The results will be presented in a scientific journal.

Importance of project Gastrostomies are commonly encumbered with minor complications, and there is a lack of evidence and guidelines on what size of gastrostomy tube that should be used. Today, local traditions or the surgeons' choice, will determine the size of the gastrostomy tube. Previously done studies are few, and to our knowledge not randomized or prospective. This study will hopefully clear the question if the size matters.

References

1. Braegger C, Decsi T, Dias JA, Hartman C, Kolacek S, Koletzko B, Koletzko S, Mihatsch W, Moreno L, Puntis J, Shamir R, Szajewska H, Turck D, van Goudoever J, ESPGHAN Committee on Nutrition (2010) Practical Approach to Paediatric Enteral Nutrition: A Comment by the ESPGHAN Committee on Nutrition. J Paediatr Gastroenterol Nutr 51(1):110-122
2. Akay B, Capizzani TR, Lee AM, Drongowski RA, Geiger JD, Hirschl RB, Mychaliska GB (2010) Gastrostomy tube placement in infants and children: is there a preferred technique? J Ped Surg 45(6):1147-1152
3. Jones VS, La Hei ER, Shun A (2007) Laparoscopic gastrostomy: the preferred method of gastrostomy in children. Pediatr Surg Int 23(11):1085-1089
4. Angsten G, Danielson J, Kassa AM, Engstrand Lilja H (2015) Outcome of laparoscopic versus open gastrostomy in children. Pediatr Sug Int 31:1067-1072
5. Merli L, De Marco EA, Fedele C, Mason EJ, Taddei A, Paradiso FV, Catania VD, Nanni L (2016) Gastrostomy Placement in children: Percutaneous Endoscopic Gastrostomy or Laparoscopic Gastrostomy? Surg Laparosc Endosc Percutan Tech 25(5):381-384
6. Danielson J, Rutqvist J, Göthberg G, Arnbjörnsson E (2018) Gastrostomi hos barn - följ nationella riktlinjer. Läkartidningen 115:E6U6
7. Franken J, Mauritz FA, Suksamanapun N, Hulsker CCC, van der See DC, van Herwaarden-Lindeboom MYA (2015) Efficacy and adverse events of laparoscopic gastrostomy placement in children: results of large cohort study. Surg Endosc 29:1545-1552
8. Townley A, Wincentak J, Krog K, Schippke J, Kingsnorth S (2017) Paediatric gastrostomy stoma complications and treatments: A rapid scoping review. J Clin Nurs 27:1369-1380
9. Jeziorczak PM, Frenette RS, Lee J, Coe SC, Aprahamian CJ (2021) Size Matters: Early Gastrostomy Tube Dislodgment in Children. J Laparoendosc Adv Surg Tech A Sep 6. doi: 10.1089/lap.2021.0352. Online ahead of print
10. Hössjer T, Göthberg G, Arnbjörnsson E, Rutqvist J, Perris F, Bartik Z, Almström M, Backman T and Danielson J (2023) Complication rate after gastrostomy placement in children can be reduced by simple surgical steps. Acta Paediatr. 2023;00;1-8. https://doi.org/10.1111/apa.16792

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for laparoscopic gastrostomy at Dep Pediatric Surgery Uppsala Akademiska University Hospital

Exclusion Criteria:

* Any specific reasons to avoid one size or the other (children who are supposed to get mixed food or a special medication that can obstruate the tube will recieve a thicker tube)

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Granuloma | 3 months postoperatively
Infection | 3 months postoperatively
Observed pain by caretakers/health care personel | 3 months postoperatively
Dislocation | 3 months postoperatively
Leakage | 3 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Barnkirurgi/Pediatric surgery, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No